CLINICAL TRIAL: NCT01800825
Title: Clindamycin to Reduce Preterm Birth in a Low Resource Setting: A Randomized Placebo-controlled Trial
Brief Title: Clindamycin to Reduce Preterm Birth in a Low Resource Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Jawaharlal Nehru Medical College (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Matthew Hoffman, Vice Chair of Department of Obstetrics and Gynecology, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Thrasher (DDD# 601465)
Record Dates: First submitted 2013-02-20; First posted 2013-02-28 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Pregnancy; Prematurity; Preterm Birth; Bacterial Vaginosis
Keywords: Pregnancy; Prematurity; Preterm birth; bacterial vaginosis
MeSH Terms: conditions — Premature Birth; Vaginosis, Bacterial | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clindamycin (Active Comparator): Clindamycin 300mg orally twice daily for five days
  Interventions: Drug: Clindamycin
- placebo (Placebo Comparator): This will be an identical placebot
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin — Clindamycin 300 mg Orally will be administered twice daily for a total of 5 days
  Other Names: Cleocin
  Arms: Clindamycin
Drug: Placebo — This will be an identical placebo comparator made of starch.
  Arms: placebo

SUMMARY:
Preterm birth has been linked to certain types of vaginal infections. The goal of this study is to determine if giving women pregnant between 13-20 weeks with an elavated vaginal pH(evidence of this type of infection)Oral Clindamycin(an antibiotic)will have a lower rate of preterm birth compared to women given a placebo(starch)

DETAILED DESCRIPTION:
The primary study objective is to definitively test whether 300 mg oral clindamycin two times per day for 5-days administered at 13-20 weeks of gestation in women with a vaginal pH≥5 reduces the incidence of preterm delivery in Karnataka, India by at least 30%. The national incidence of gestation <37 weeks in India is 14.5%, was 18% in the study area in 2011 and was 20% among women with vaginal pH≥5 in the recently completed Jawaharlal Nehru Medical Collage (JNMC) hospital-based study of clindamycin to reduce preterm birth. Using a two tailed test, α=0.05, 1-β=80%, a 17.5% rate of prematurity in women with vaginal pH≥5, a 2.5% refusal and a 7.5% loss to follow-up, assuming 86% of women presenting for antenatal care are 13-20 weeks gestation and 1% otherwise ineligible, and a multiple comparisons adjustment, 1,726 women, half in the clindamycin and half in the placebo group, need to be enrolled to test the primary hypothesis. The effects of clindamycin on spontaneous preterm birth, miscarriage, low birthweight (LBW), neonatal mortality (NMR), maternal and neonatal complications through 42 days postpartum, the utility of vaginal pH≥5 to identify women at risk for preterm delivery and the costs of preterm birth prevented by oral clindamycin treatment and compliance with the 5-day treatment regimen will also be assessed. This will be the first investigation to test whether oral clindamycin prevents preterm birth in a community-based, developing country setting, where most global newborn deaths occur.

ELIGIBILITY:
Inclusion Criteria:

* Women with a singleton Intrauterine pregnancy between 13-20 weeks
* Maternal age of 18 or older or if < 18 assent of the women's parent/guardian
* Vaginal PH > 5.0

Exclusion Criteria:

* Use of antibiotics within the 14 days prior to randomization
* Known sensitivity to antibiotics
* Uterine anomalies
* Major fetal anomalies
* Medical conditions that may result in iatrogenic prematurity(e.g.diabetes, Lupus, Hypertension)

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1726 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Preterm birth prior to 37 weeks | Time of birth
  Preterm birth prior to 37 weeks

SECONDARY OUTCOMES:
Preterm birth prior to 34 weeks | Time of birth
  Preterm birth prior to 34 weeks
Late Miscarriage | Time of delivery
  miscarriage between 16-20 weeks
Low Birth weight | Time of delivery
  Birth Weight< 2500 gm
Very Low birth Weight | Time of delivery
  Very Low birth Weight is birthweight <1500gm
Neonatal complications through 42 days after delivery | 42 days post delivery
  Neonatal complications through 42 days after delivery (to assess benefit or no harm)
Maternal complications through 42 days postpartum | 42 days post delivery
  Maternal complications through 42 days postpartum (to assess benefit or no harm)
The utility of vaginal pH tests for identification of women at elevated risk for preterm delivery | Time of delivery
  The utility of vaginal pH tests for identification of women at elevated risk for preterm delivery

OTHER OUTCOMES:
neonatal mortality | Time of delivery
  neonatal mortality
maternal and neonatal complications through 42 days postpartum, | 42 days postpartum
  maternal and neonatal complications through 42 days postpartum,
Incremental cost of preventing preterm birth | 42 days postpartum
  Determine the costs of preventing preterm birth

CONTACTS AND LOCATIONS:
Overall Officials: Matthew K Hoffman, MD MPH, Principal Investigator — Christiana Care Health Services
Locations (1):
- Jawaharlal Nehru Medical College, Belagavi, Karnataka, India

REFERENCES:
- [Background] Lamont RF, Nhan-Chang CL, Sobel JD, Workowski K, Conde-Agudelo A, Romero R. Treatment of abnormal vaginal flora in early pregnancy with clindamycin for the prevention of spontaneous preterm birth: a systematic review and metaanalysis. Am J Obstet Gynecol. 2011 Sep;205(3):177-90. doi: 10.1016/j.ajog.2011.03.047. Epub 2011 Apr 2. PMID 22071048
- [Background] Ugwumadu A, Manyonda I, Reid F, Hay P. Effect of early oral clindamycin on late miscarriage and preterm delivery in asymptomatic women with abnormal vaginal flora and bacterial vaginosis: a randomised controlled trial. Lancet. 2003 Mar 22;361(9362):983-8. doi: 10.1016/S0140-6736(03)12823-1. PMID 12660054
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Lawn JE, Blencowe H, Pattinson R, Cousens S, Kumar R, Ibiebele I, Gardosi J, Day LT, Stanton C; Lancet's Stillbirths Series steering committee. Stillbirths: Where? When? Why? How to make the data count? Lancet. 2011 Apr 23;377(9775):1448-63. doi: 10.1016/S0140-6736(10)62187-3. Epub 2011 Apr 13. PMID 21496911
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Friese K. The role of infection in preterm labour. BJOG. 2003 Apr;110(Suppl 20):52-4. doi: 10.1016/s1470-0328(03)00025-9. PMID 12763112
- [Background] Hauth JC, Goldenberg RL, Andrews WW, DuBard MB, Copper RL. Reduced incidence of preterm delivery with metronidazole and erythromycin in women with bacterial vaginosis. N Engl J Med. 1995 Dec 28;333(26):1732-6. doi: 10.1056/NEJM199512283332603. PMID 7491136
- [Background] Hutzal CE, Boyle EM, Kenyon SL, Nash JV, Winsor S, Taylor DJ, Kirpalani H. Use of antibiotics for the treatment of preterm parturition and prevention of neonatal morbidity: a metaanalysis. Am J Obstet Gynecol. 2008 Dec;199(6):620.e1-8. doi: 10.1016/j.ajog.2008.07.008. Epub 2008 Oct 30. PMID 18973872
- [Background] McDonald HM, Brocklehurst P, Gordon A. Antibiotics for treating bacterial vaginosis in pregnancy. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD000262. doi: 10.1002/14651858.CD000262.pub3. PMID 17253447
- [Background] Joesoef MR, Hillier SL, Wiknjosastro G, Sumampouw H, Linnan M, Norojono W, Idajadi A, Utomo B. Intravaginal clindamycin treatment for bacterial vaginosis: effects on preterm delivery and low birth weight. Am J Obstet Gynecol. 1995 Nov;173(5):1527-31. doi: 10.1016/0002-9378(95)90644-4. PMID 7503196
- [Background] Lamont RF. Antibiotics for the prevention of preterm birth. N Engl J Med. 2000 Feb 24;342(8):581-3. doi: 10.1056/NEJM200002243420810. No abstract available. PMID 10684919
- [Background] Guaschino S, Ricci E, Franchi M, Frate GD, Tibaldi C, Santo DD, Ghezzi F, Benedetto C, Seta FD, Parazzini F. Treatment of asymptomatic bacterial vaginosis to prevent pre-term delivery: a randomised trial. Eur J Obstet Gynecol Reprod Biol. 2003 Oct 10;110(2):149-52. doi: 10.1016/s0301-2115(03)00107-6. PMID 12969574
- [Background] Kurkinen-Raty M, Vuopala S, Koskela M, Kekki M, Kurki T, Paavonen J, Jouppila P. A randomised controlled trial of vaginal clindamycin for early pregnancy bacterial vaginosis. BJOG. 2000 Nov;107(11):1427-32. doi: 10.1111/j.1471-0528.2000.tb11660.x. PMID 11117774
- [Background] Kekki M, Kurki T, Pelkonen J, Kurkinen-Raty M, Cacciatore B, Paavonen J. Vaginal clindamycin in preventing preterm birth and peripartal infections in asymptomatic women with bacterial vaginosis: a randomized, controlled trial. Obstet Gynecol. 2001 May;97(5 Pt 1):643-8. doi: 10.1016/s0029-7844(01)01321-7. PMID 11339909
- [Background] Morency AM, Bujold E. The effect of second-trimester antibiotic therapy on the rate of preterm birth. J Obstet Gynaecol Can. 2007 Jan;29(1):35-44. doi: 10.1016/s1701-2163(16)32350-7. PMID 17346476
- See also: Thrasher Foundation — http://www.thrasherresearch.org/